CLINICAL TRIAL: NCT02545400
Title: Quantification of Side Effects During Dual or Triple Therapy for Chronic Hepatitis C
Brief Title: Quantification of Side Effects During Hepatitis C Therapy
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: HCV-side effects
Record Dates: First submitted 2015-07-29; First posted 2015-09-10 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to assess the frequency and severity of adverse events during Hepatitis C therapy with or without first generation protease inhibitors.

DETAILED DESCRIPTION:
Hepatitis C Virus infection is one of the main causes of chronic liver disease worldwide with current estimates of approximately 130 - 210 million individuals (according to 3% of the world population) chronically infected with the hepatitis C virus. However, hepatitis C virus infections are among the most common causes leading to chronic hepatitis, liver cirrhosis and liver related death worldwide.

The current standard of care is a combination of pegylated Interferon and Ribavirin (dual-therapy). Since 2011, direct-acting antiviral drugs inhibiting viral protease are approved as an addition to the standard therapy (triple-therapy).

The occurrence of adverse events as well as their severity generally depends on the therapy regimen and is influenced by type and dosage of medications.

Most common adverse events (affects up to 95% of patients) are fever, fatigue, headache, nausea, arthralgia, depression, skin reactions, neutropenia, and anemia.

A more frequent occurrence of adverse events with triple-therapy compared to dual- therapy has become clear since it's introduction, particularly with regard to anemia, neutropenia, gastrointestinal discomfort, fatigue, dysgeusia, and skin reactions. How- ever, there is accumulating evidence for a more often appearance of infections and/or infestations in patients receiving triple-therapy.

The medical consequence from adverse events is a reduction of quality of life and consecutively the loss of antiviral therapy adherence. Thus, early recognition and immediate treatment of adverse events are crucial aspects in the success of antiviral treatment.

Aim of this study is to quantify reported adverse events with respect to therapy reg- imen (dual-therapy vs. triple-therapy) in patients who are treated at the Department of Internal Medicine, Division of Gastroenterology and Hepatology at the Medical University Graz. Furthermore, a detailed review of international treatment recommendations, as well as an analysis of possible predictor parameters for the appearance of adverse events and treatment success is done.

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis C
* Indication for a hepatitis C therapy

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C undergoing therapy with pegylated interferon and ribavirin +/- a firstgeneration protease inhibitor
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
frequency of adverse events | on average 24 weeks
  reported adverse events

SECONDARY OUTCOMES:
type of adverse events | on average 24 weeks
  reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Stadlbauer, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria

REFERENCES:
- [Derived] Spindelboeck W, Horvath A, Tawdrous M, Schmerbock B, Zettel G, Posch A, Streit A, Jurse P, Lemesch S, Horn M, Wuensch G, Stiegler P, Stauber RE, Leber B, Stadlbauer V. Triple Therapy with First Generation Protease Inhibitors for Hepatitis C Markedly Impairs Function of Neutrophil Granulocytes. PLoS One. 2016 Mar 3;11(3):e0150299. doi: 10.1371/journal.pone.0150299. eCollection 2016. PMID 26938078